CLINICAL TRIAL: NCT06913127
Title: Does High-intensity Exercise Lead to Better Functional Outcomes Early After Stroke in an Inpatient Rehabilitation Setting?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mah Shi Min (Other)
Responsible Party: Sponsor-Investigator, Mah Shi Min, Senior Principal Physiotherapist, Sengkang General Hospital
Organization: Sengkang General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-3187
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; High-intensity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High intensity exercise (Experimental): High intensity exercise: 60-84% HRR (heart rate reserve) or RPE (rate of perceived exertion) 14-16 HR max for people on beta-blockers: 164- (0.7 x Age) HR max for people not on beta-blockers: 206.9 -(0.67 x Age)
  Interventions: Other: High intensity exercise post stroke
- Low intensity exercise (Active Comparator): Low intensity exercise: 59% HRR and below (heart rate reserve) or RPE (rate of perceived exertion) 13 and below HR max for people on beta-blockers: 164- (0.7 x Age) HR max for people not on beta-blockers: 206.9 -(0.67 x Age)
  Interventions: Other: High intensity exercise post stroke

INTERVENTIONS:
Other: High intensity exercise post stroke — The patients are all admitted with an acute/ subacute stroke in an inpatient rehabilitation ward. They are randomized into a high intensity exercise or a low intensity exercise group that will last for 20 consecutive sessions. At the end of the experimental period, outcomes including functional outcomes, questionnaires, physical activity and fNIRS (functional near infrared spectroscopy) measurements will be compared between the two groups.

SUMMARY:
The purpose of this study is to find out the effectiveness of high intensity exercise (HIE) early after stroke, this study is hoping to recruit 36 participants in total and will be analysing pre- and post- outcomes of patients in a high intensity exercise intervention, as compared to a lower intensity exercise programme. Participants will be randomly assigned to either the high or low intensity exercise programme, and receiving the assigned intervention for 2 weeks. Both groups in the study will be subjected to same post-stroke functional and locomotion training as part of their physiotherapy intervention, but at different intensities. This ranges from body weight supported training, to treadmill training, to robotics walking and functional training (including overground walking/ stepping and cardiorespiratory fitness training), as per conventional post-stroke rehabilitation.

The high intensity experimental group will undergo high-intensity exercise (HIE) training defined by 60-84% (heart rate reserve), or RPE (rate of perceived exertion) Borg 14-16, while the low intensity control group will undergo lower intensity training defined by HRR 59% and below, or RPE Borg 13 and below.

Measurements will be taken from assessments at pre- and post- interventions will be analysed and compared between the two groups to find out which intervention programme is more effective for patients early after stroke. These assessments include functional outcomes such as walking speed, chair rise test and also a neurobiological measure looking at levels of cortical activation called the functional near infrared spectroscopy (fNIRS) which is measured via a non-invasive cap that you wear on. The participants will be expected to don on the fNIRS device for a total of 15-30 minutes, and an average of 3 sets of 30-seconds measurements during their walking assessment will be taken.

DETAILED DESCRIPTION:
Research participants are warded in an inpatient rehabilitation unit during the duration of the intervention. Prior to the enrolment of the patients into the study, the neurologist/ neurosurgeon or primary physician will be consulted of the suitability of their patient in performing high intensity exercise during their physiotherapy sessions as part of this trial. The exercise intensity parameters that the participants will be subjected to, will also be informed to the medical team before the start of the exercise intervention, with clarifications on any additional precautions or parameters to adhere to, to ensure that the participants are fit and safe to be recruited into this exercise trial. After enrolment, participants will be randomized into experimental and control group by concealed allocation by a neutral party.

Pre- and post- intervention outcomes will be measured by blinded therapists, and compared between groups; the outcome measurements include Functional Independence Measure (FIM), Berg Balance Scale (BBS), Mobility Scale for Acute Stroke (MSAS), Five time Sit to Stand Test (5 STS), gait speed, fatigue severity scale (FSS), and motivation in stroke patients for rehabilitation (MORE) scale. The outcomes will be recorded and analyzed to examine the effectiveness of high intensity exercise (HIE) post stroke. Functional near infrared spectroscopy (fNIRS), a non-invasive optical brain monitoring device, will be donned on during walking tests to monitor and compare the cortical activity in both groups. An average of 3 sets of 30-second measurements with the fNIRS will be taken during walking, the participant will be expected to wear the device for 15-30 minutes. Physical activity tracking via number of steps/ day and activity log will be used to monitor the effects of the interventions on the patients' activity levels while warded.

Exercise intervention: All patients will be subjected to standard post-stroke functional and locomotion training as part of their physiotherapy intervention. This ranges from body weight supported training, to treadmill training, to robotics walking and functional training (including overground walking/ stepping and cardiorespiratory fitness training), as per conventional post-stroke rehabilitation. Both groups will undergo the same training as described above, prescribed by their physiotherapist; the only difference is the intensity of the exercise. The experimental group will undergo high-intensity exercise (HIE) training defined by 60- 84% HRR (heart rate reserve) or RPE (rate of perceived exertion) Borg Scale 14-16, while the control group will undergo lower intensity training defined by HRR 59% and below, or RPE Borg 13 and below.

Safety monitoring: Prior to start of exercise interventions, patients will be asked if they feel unwell or present with any symptoms that are of concern, their vitals (HR, BP, RR and spO2) will be taken. Throughout the session, HR will be monitored and spO2, BP and RR will be taken every 2-5 minutes to ensure that they are within safe limits. Immediately after exercise and post session, patients will be asked for their symptoms and vitals will again be taken. All vitals monitoring will be recorded, and the attending physiotherapist or patient is able to stop the intervention at any time if they feel that the physiological measures/ responses are not within safe limits for the intervention to continue.

In accordance to literature review of similar topics, post stroke exercise intensity in this study will be definedas such: Target HR= Target HRR % x (HR max- HR resting)+ HR resting HR max for people not on beta-blockers= 206.9 - (0.67 x Age) HR max for people on beta-blockers: 164 - (0.7 x Age) High intensity exercise: 60-84% HRR OR RPE Borg 14-16

A medical record review of the patients enrolled into the study will be conducted where patient characteristics, including demographic data, type of stroke, site of lesion, stroke severity (NIHSS), nature of impairments, cognitive level (MOCA) and use of medications, premorbid and pre-rehabilitation functional status will be documented. Functional outcome measures will be evaluated at the start and end of the intervention period (i.e. after 2 weeks, 10 days bidaily- 20 sessions) of inpatient rehabilitation training.

Data analysis: Statistical analysis will be conducted to examine the difference in outcomes between the experimental and control groups. If the hypotheses of this study that HIE is more effective in improving outcomes as compared to low intensity is proven to be accurate, this will have clinical implications in provision of high quality evidence based care as it contributes to advocating for HIE to implemented in standard stroke care in the acute inpatient rehabilitation centres in Singapore, and worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted for acute ischaemic or haemorrhagic stroke and requiring inpatient rehabilitation for stroke
2. First-ever, single, unilateral stroke
3. Aged 21-99 years old
4. Able to walk 10m overground with minimal or moderate physical assistance
5. Cleared by physician to be medically stable to participate in high intensity exercise (HIE)
6. Participants have to be warded for inpatient rehabilitation for at least 10 consecutive weekdays

Exclusion Criteria:

1. Any central or peripheral nervous system or orthopedic injury that may limit ambulation or exercise
2. Uncontrolled cardiorespiratory disease
3. Inability to follow 3 steps commands
4. Patient unable to give consent for the study
5. Patient who is assessed unsuitable to don on the medical device fNIRS (eg patients who had undergone craniectomy and cranioplasty)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure | At enrollment and at end of treatment at 2 weeks
  The FIM (Functional Independence Measure) score is a standardized tool used to assess a patient's functional independence during rehabilitation, with scores ranging from 18 to 126, where higher scores indicate greater independence.
Berg Balance Scale | At enrollment and at end of treatment at 2 weeks
  The Berg balance scale (BBS) is widely used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a set of 14 simple balance related tasks, ranging from standing up from a sitting position to standing on one foot, and takes approximately 20 minutes to complete. Each item is scored 0 to 4, resulting in a total score ranging from 0 to 56, where higher scores indicate better balance.
Mobility Scale for Acute Stroke (MSAS) | At enrollment and at end of treatment at 2 weeks
  The Mobility Scale for Acute Stroke (MSAS) is a unidimensional instrument that produces a single aggregate score from 6 basic mobility activities that correspond with the range of abilities seen in people with acute stroke. The 6 activities are scored using a 6-point scale, with total scores ranging from 6 to 36, where a lower score indicates more assistance is required.
Five Times Sit to Stand Test | At enrollment and at end of treatment at 2 weeks
  The Five Times Sit to Stand Test (5x Sit-To-Stand Test) is commonly abbreviated as 5XSST. It's used to asses functional lower limbs strength, transitional movements, balance, and fall risk.
Gait Speed | At enrollment and at end of treatment at 2 weeks
  Gait speed, or walking speed, is a measure of how quickly someone can walk a specified distance, calculated by dividing the distance by the time taken, and is often expressed in meters per second (m/s). It's a valuable indicator of functional ability and can be used to assess fall risk.
Fatigue Severity Scale | At enrollment and at end of treatment at 2 weeks
  The Fatigue Severity Scale (FSS) is a 9-item questionnaire used to measure the severity of fatigue and its impact on daily life, with higher scores indicating greater fatigue.
Motivation in stroke patients for rehabilitation (MORE) scale | At enrollment and at end of treatment at 2 weeks
  The MORE scale, or Motivation in stroke patients for rehabilitation scale, is a 17-item tool developed to assess stroke patients' motivation for rehabilitation, exploring both intrinsic and extrinsic factors, with higher scores indicating higher motivation.

SECONDARY OUTCOMES:
Steps per day | Daily, throughout 2-weeks intervention
  Steps per day will be tracked, and recorded.
Physical Activity Log | Daily, throughout 2-weeks intervention
  Patients will record the physical activity he/ she performed that day, as well as how he/ she felt, and any additional comments.

OTHER OUTCOMES:
fNIRS (functional near-infrared spectroscopy) during walking tasks | At enrollment and at end of treatment at 2 weeks
  fNIRS (functional near-infrared spectroscopy) is a non-invasive neuroimaging technique that uses near-infrared light to measure changes in blood oxygenation in the brain, providing an indirect measure of brain activity. fNIRS will be used in the 3 sets of 30s walk test, and measured pre and post- intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
The data is intended to be shared at conference, and yet to be published.

REFERENCES:
- [Background] Robertson AD, Crane DE, Rajab AS, Swardfager W, Marzolini S, Shirzadi Z, Middleton LE, MacIntosh BJ. Exercise intensity modulates the change in cerebral blood flow following aerobic exercise in chronic stroke. Exp Brain Res. 2015 Aug;233(8):2467-75. doi: 10.1007/s00221-015-4317-6. Epub 2015 May 24. PMID 26003127
- [Background] Globas C, Becker C, Cerny J, Lam JM, Lindemann U, Forrester LW, Macko RF, Luft AR. Chronic stroke survivors benefit from high-intensity aerobic treadmill exercise: a randomized control trial. Neurorehabil Neural Repair. 2012 Jan;26(1):85-95. doi: 10.1177/1545968311418675. Epub 2011 Sep 1. PMID 21885867
- [Background] Chan, C. Y., Mullen, M., Burrows, J., Kerr, I., Petrunia, C., Dawson, A., & Feehan, L. (2015). Targeted dischargeplanning for stroke clients in high intensity rehabilitation settings is associated with a notable reductioninlength of stay. International Journal of Stroke, 10, 78-78.
- [Background] Askim T, Dahl AE, Aamot IL, Hokstad A, Helbostad J, Indredavik B. High-intensity aerobic interval training for patients 3-9 months after stroke: a feasibility study. Physiother Res Int. 2014 Sep;19(3):129-39. doi: 10.1002/pri.1573. Epub 2013 Dec 4. PMID 24375978